CLINICAL TRIAL: NCT07188558
Title: A Phase 3 Randomized Controlled Trial of Rondecabtagene Autoleucel , an Autologous, Dual-targeting CD19/CD20 CAR T-Cell Product Candidate, Vs. Investigator's Choice of CD19 CAR T-Cell Therapy in Patients With Relapsed or Refractory Large B-Cell Lymphoma in the Second-line Setting
Brief Title: A Study to Investigate Ronde-cel Versus Investigator's Choice CD19 CAR T-Cell Therapy
Acronym: PiNACLE-H2H
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lyell Immunopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYL314-102
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Large B-cell Lymphoma; Lymphoma, B-Cell; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Non-Hodgkin Lymphoma Refractory/ Relapsed; Diffuse Large B Cell Lymphoma (DLBCL); Diffuse Large B Cell Lymphoma Refractory; Diffuse Large B Cell Lymphoma Relapsed
Keywords: Lymphoma; Non-Hodgkin Lymphoma; CAR T-Cell Therapy; CD19; CD19/CD20; Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rondecabtagene autoleucel (Experimental)
  Interventions: Biological: rondecabtagene autoleucel
- Investigator's Choice CD19 (Active Comparator): axicabtagene ciloleucel, lisocabtagene maraleucel
  Interventions: Biological: axicabtagene ciloleucel; Biological: lisocabtagene maraleucel

INTERVENTIONS:
Biological: rondecabtagene autoleucel — An autologous, dual-targeting CD19/20 CAR T-cell candidate.
  Other Names: LYL314
  Arms: Rondecabtagene autoleucel
Biological: axicabtagene ciloleucel — An autologous CD19 CAR T-cell therapy
  Other Names: Yescarta; axi-cel
  Arms: Investigator's Choice CD19
Biological: lisocabtagene maraleucel — An autologous CD19 CAR T-cell therapy
  Other Names: Breyanzi; liso-cel
  Arms: Investigator's Choice CD19

SUMMARY:
This Phase 3 study compares rondecabtagene autoleucel (ronde-cel), a dual-targeting CD19/CD20 CAR T-cell therapy, with investigator's choice of CD19 CAR T-cell therapy in patients with relapsed or refractory large B-cell lymphoma in the second-line setting.

DETAILED DESCRIPTION:
PiNACLE-H2H is a Phase 3 randomized controlled trial comparing the efficacy and safety of rondecabtagene autoleucel (ronde-cel, formerly known as LYL314) against the currently approved cluster of differentiation (CD)19 chimeric antigen receptor (CAR) T-cell therapies (axicabtagene ciloleucel [axi-cel] or lisocabtagene maraleucel [liso-cel]), in patients with aggressive LBCL that has relapsed or is refractory to first-line anti-CD20 antibody and anthracycline-containing chemotherapy.

Patients will be randomized (1:1) before leukapheresis to receive either:

* Ronde-cel; or
* Investigator's choice of axi-cel or liso-cel

Most patients who receive currently approved CD19-directed CAR T-cell therapies, including axi-cel and liso-cel, still experience progressive disease, often due to mechanisms such as CD19 antigen loss or T-cell exhaustion.

Ronde-cel is a novel, autologous, dual-targeting CD19/CD20 CAR T-cell product candidate enriched for CD62L-positive naïve and central memory T cells, which are associated with enhanced proliferation capacity and persistence. Ronde-cel is an "OR"-gated CAR construct that can fully activate upon recognition of either CD19 or CD20, aiming to improve durability of response despite antigen heterogeneity.

Approximately 400 participants will be enrolled. CAR T-cell therapy in both arms will be administered as a single intravenous infusion following fludarabine and cyclophosphamide lymphodepletion. Participants will be followed for 3 years for safety and efficacy, with long-term follow-up extending to 15 years.

ELIGIBILITY:
Key Inclusion Criteria:

1. CAR T cell naïve and eligible to receive a CD19 CART-cell therapy
2. Histologically confirmed large B-cell lymphoma, including the following types defined by (WHO 2022) or International Consensus Classification (2022)

   * Diffuse large B-cell lymphoma (DLBCL)
   * Transformations of indolent B-cell lymphomas (excluding Richter's transformation)
   * DLBCL/High-grade B-cell lymphoma (HGBCL) with MYC and BCL2 rearrangements
   * High-grade B-cell lymphoma (HGBCL) not otherwise specified (HGBCL NOS)
   * Primary mediastinal large B-cell lymphoma (PMBCL)
   * Grade 3B follicular lymphoma/large cell follicular lymphoma (FL3B)
3. Relapsed or refractory disease after anti-CD20 antibody and anthracycline-containing first-line chemoimmunotherapy
4. Measurable disease by presence of [18F]-fluorodeoxyglucose PET/CT positive lesion during Screening per Lugano Criteria
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Adequate hematological, renal, hepatic, pulmonary, and cardiac function

Key Exclusion Criteria:

1. Patients ineligible to receive CD19 CAR T-cell therapy
2. Primary CNS lymphoma
3. Patients with primary cutaneous LBCL, human herpes virus-8 positive lymphoma, Burkitt lymphoma, T cell histiocyte-rich lymphoma, or transformation from chronic lymphocytic leukemia/small lymphocytic lymphoma (Richter's transformation)
4. Patients with prior history of malignancy, other than aggressive relapsed or refractory LBCL, unless the patient has been free of the disease for ≥ 2 years
5. Patients with uncontrolled systemic fungal, bacterial, viral, or other infection (including tuberculosis) despite appropriate antibiotics or other treatment
6. Active autoimmune disease requiring ongoing systemic immunosuppressive therapy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 36 months
  The time interval from treatment initiation until the occurrence of a specific event of interest.

SECONDARY OUTCOMES:
Overall Response Rate | 36 months
  Best Overall Response per Lugano Criteria
Complete Response Rate | 36 months
  Complete Response per Lugano Criteria
Progression Free Survial | 36 months
  The length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Overall Survival | 6 years
  The length of time from either the date of diagnosis or the start of treatment for a disease, that patients diagnosed with the disease, are still alive.
Incidence and severity adverse events | 36 months
  To assess safety defined as type and frequency of AEs, serious adverse events (SAEs), and laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Honor Health, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of Colorado, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - AdventHealth, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville Health, Louisville, Kentucky
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center (UNMC), Omaha, Nebraska
  - Hackensack, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Oncology Hematology Care Clinical Trials, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinical Taussig Cancer Center, Cleveland, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - University of Texas Southwestern Medical Center, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Swedish Cancer Institute, Seattle, Washington